CLINICAL TRIAL: NCT07302464
Title: Effect of Sodium Glucose Co-Transporter 2 Inhibitors on Estimated Glomerular Filtration Rate in Diabetic Versus Non-Diabetic Chronic Kidney Disease Patients
Brief Title: Sodium Glucose Co-Transporter 2 Inhibitors on Estimated Glomerular Filtration Rate in Diabetic Versus Non-Diabetic Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf Hassan, Assistant Professor of Internal Medicine and Nephrology, Faculty of Medicine, Ain shams University, Cairo, Egypt, Ain Shams University
Other Study IDs: FMASU MS 603/2024
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Sodium Glucose Co-Transporter 2 Inhibitors; Estimated Glomerular Filtration Rate; Diabetes; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Chronic kidney disease (CKD) participants with type 2 diabetes mellitus (T2DM)
  Interventions: Other: Sodium Glucose Co-Transporter 2 Inhibitors
- Control group: Chronic kidney disease (CKD) participants without diabetes mellitus
  Interventions: Other: Sodium Glucose Co-Transporter 2 Inhibitors

INTERVENTIONS:
Other: Sodium Glucose Co-Transporter 2 Inhibitors — All candidates start therapy with sodium glucose co-transporter 2 (SGLT2) inhibitors with a dose of 10mg daily Dapagliflozin for 6 months

SUMMARY:
The work aimed to compare the effects of Sodium-glucose co-transporter-2 (SGLT2) inhibitors on glomerular filtration rate (GFR) in patients with diabetic chronic kidney disease (CKD) and non-diabetic CKD.

DETAILED DESCRIPTION:
Glucose reabsorption is mediated by the sodium-glucose cotransporter (SGLT) 2, which reabsorbs 90% of glucose, and SGLT1, which reabsorbs the remaining 10%.

The relationship between hyperglycaemia and the development of renal disease is complex. Hyperglycaemia-induced complications are mediated by several metabolic pathways, among which accumulation of Advanced Glycation End-products with abnormalities of the glycosylation of macromolecules and increased glucose flux through the polyol pathway seem to be the most important.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Chronic kidney disease (CKD) participants with stages 3 and 4.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus (DM).
* Patients with decompensated Chronic liver disease.
* Patients with uncontrolled hypertension.
* Patients with blood pressure (BP) > 110/70.
* Patients already on the same medication (Sodium Glucose Co-Transporter 2 Inhibitors).
* Patients with a history of recurrent or recent urinary tract infection (UTI).
* Patients with glycated hemoglobin (HbA1c) ≤10.
* Adult polycystic kidney disease.
* All patients on immunosuppressive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This case-control study was done on 60 adult chronic kidney disease (CKD) individuals with stage 3 and 4 (eGFR>_20ml/min/1.73 m2) according to KIDGO classification at Ain Shams University Hospitals, Cairo, Egypt.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in the estimated glomerular filtration rate | 6 months post-procedure
  Change in the estimated glomerular filtration rate (eGFR) was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.